CLINICAL TRIAL: NCT03832088
Title: Sarcopenia And Balance In Postmenopausal Osteoporosis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Medeniyet University (Other)
Responsible Party: Principal Investigator, Bilinç Doğruöz Karatekin, MD, Research Assistant of PMR, Istanbul Medeniyet University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: MedeniyetOP
Record Dates: First submitted 2019-02-02; First posted 2019-02-06 (Actual); Last update posted 2019-02-21 (Actual); Status verified 2019-02

CONDITIONS: Osteoporosis, Postmenopausal; Balance; Distorted; Sarcopenia
Keywords: osteoporosis; sarcopenia; balance disorder
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Sarcopenia; Osteoporosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- postmenopausal osteoporosis (Experimental): Postmenopausal osteoporotic patients evaluated for sarcopenia and balance disorders
  Interventions: Diagnostic Test: Berg Balance Scale; Diagnostic Test: Timed Up and Go Test; Diagnostic Test: Jamar hand dynamometer; Diagnostic Test: Calf circumference

INTERVENTIONS:
Diagnostic Test: Berg Balance Scale — Berg Balance Scale performed for balance disorder
Diagnostic Test: Timed Up and Go Test — Timed Up and Go Test for walking speed
Diagnostic Test: Jamar hand dynamometer — Jamar hand dynamometer for grip strength which correlates with muscle strength of patient
Diagnostic Test: Calf circumference — Calf circumference for muscle mass evaluation. Calf circumference is an anthropometric measurement which correlates with muscle mass.

SUMMARY:
The study was performed on 53 postmenopausal osteoporosis patients who presented to our osteoporosis outpatient clinic. Following written informed consent, patients were evaluated for sarcopenia according to the sarcopenia algorithm proposed by the European Working Group on Sarcopenia in Older People (EWGSOP). Algorithm parameters were walking speed, muscle strength and muscle mass measurements. We used Timed Up and Go Test (TUG) for evaluation of walking speed, Jamar Hand Dynamometer for muscle strength assessment, and calf circumference for muscle mass measurement. Balances of the patients were evaluated with Berg Balance Scale (BBS) and functional skills were evaluated with the Timed Up and Go Test (TUG). Other clinical parameters (age, body mass index (BMI), 25OHvitD level, menopause age, fall within the last year, fracture history, history of fracture in mother) were questioned.

DETAILED DESCRIPTION:
The study was performed on 53 postmenopausal osteoporosis patients who presented to our osteoporosis outpatient clinic. Following written informed consent, patients were evaluated for sarcopenia according to the sarcopenia algorithm proposed by the European Working Group on Sarcopenia in Older People (EWGSOP). Algorithm parameters were walking speed, muscle strength and muscle mass measurements. We used Timed Up and Go Test (TUG) for evaluation of walking speed, Jamar Hand Dynamometer for muscle strength assessment, and calf circumference for muscle mass measurement. Balances of the patients were evaluated with Berg Balance Scale (BBS) and functional skills were evaluated with the Timed Up and Go Test (TUG). Other clinical parameters (age, body mass index (BMI), 25OHvitD level, menopause age, fall within the last year, fracture history, history of fracture in mother) were questioned. SPSS 22.0 program will be used for statistical evaluation and correlation analysis will be done.

ELIGIBILITY:
Inclusion Criteria:

* Having postmenopausal osteoporosis
* No other disease that can cause balance disorder
* Volunteer participation in the study

Exclusion Criteria:

* To have a disease that will cause balance disorder,
* Having understanding problem to prevent communication with the patient,
* The lack of motor function to the balance device.

Min Age: 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Postmenopausal osteoporotic patients
Enrollment: 53 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
sarcopenia in postmenopausal osteoporotic patients | 6 months
  sarcopenia evaluated according to EWGSOP algorithm which includes walking speed, muscle strength and muscle mass measures
balance disorder in postmenopausal osteoporotic patients | 6 months
  balance evaluated by Berg Balance Scale ( 0-56 scored scale , bigger score indicates better balance, scores under 41 indicates bigger risk of falling )

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medeniyet University Faculty of Medicine, Physical Therapy and Rehabilitation Department, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided